CLINICAL TRIAL: NCT01605760
Title: House Dust Mite Sublingual Immunotherapy: a Double-blind, Placebo Control Study in Elderly Patients.
Brief Title: House Dust Mite SLIT in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Andrzej Bozek, Medical Doctor, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 657898/2008
Record Dates: First submitted 2012-05-17; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Allergic Rhinitis
Keywords: immunotherapy; elderly
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non immunotherapy treatment (No Intervention)
  Interventions: Drug: immunotherapy Staloral
- sublingual immunotherapy course (Active Comparator)
  Interventions: Drug: immunotherapy Staloral

INTERVENTIONS:
Drug: immunotherapy Staloral — Staloral (R) 300 is a sublingual solution of allergen extracts for allergen immunotherapy. During a 16 day incrementally increasing dose period, patients took daily increasing doses period, patients took 1-8 drops of the 100 IR/ml extract during the first 8 days. Then, on days 9-16, patients took 1-8 drops of the 300 IR/ml extract. Next, patients received maintenance treatment consisting of five applications of eight drops (equivalent to 0.5 mL) of 300 IR/mL extract five times a week. The mean duration of the treatment was 28.2 months (range: 3-36 months).

SUMMARY:
The safety and efficacy of specific sublingual immunotherapy for house dust mite allergens in patients over 60 years of age with allergic rhinitis and a confirmed allergy to house dust mites were the focus of the stu First, 111 patients, ages 60-75 years, with allergic rhinitis and with a confirmed allergy to D. pteronyssinus and D. farinae by the use of skin prick tests, serum-specific IgE and nasal provocation tests were included. Patients were individually randomised to groups: active or placebo using a double-blind method. A total of 51 subjects in the sublingual allergen-specific immunotherapy (SLIT) group (Staloral 300R, Stallergens, France) and 57 in the placebo group were monitored for three years. The patients had to record on a diary card whenever they used anti-allergic medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with allergic rhinitis who fulfilled the ARIA criterion and had a positive skin prick test (SPT), were positive for specific immunoglobulin E (sIgE) and had positive nasal provocation tests (NPTs) by Dermatophagoides pteronyssinus (Der p) and Dermatophagoides farinae (Der f) were included in the study

Exclusion Criteria:

* Patients with any of the following characteristics were excluded:

  * hypersensitivity to other allergens,
  * non-allergic rhinitis (especially senile or vasomotor rhinitis) or
  * severe non-stable diseases (especially bronchial asthma). However, stable coronary disease, diabetes, arterial hypertension and well-controlled, mild or atopic bronchial asthma were permitted.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse event during immunotherapy | three year
  Safety assessment of sublingual immunotherapy on the basis of the monitoring clinical adverse events during treatment by the use of a patient diary and medical examination.

SECONDARY OUTCOMES:
Change from baseline of nasal symptoms after immunotherapy | three year
  Assessment of reducing the need for symptom-targeted drugs, primarily antihistamines and reducing of nasal symptoms during treatment in study patients (diary monitoring).

CONTACTS AND LOCATIONS:
Locations (1):
- Allergology Outpatient Clinic, Zabrze, Poland

REFERENCES:
- [Derived] Bozek A, Starczewska-Dymek L, Jarzab J. Prolonged effect of allergen sublingual immunotherapy for house dust mites in elderly patients. Ann Allergy Asthma Immunol. 2017 Jul;119(1):77-82. doi: 10.1016/j.anai.2017.05.012. PMID 28668244
- [Derived] Bozek A, Ignasiak B, Filipowska B, Jarzab J. House dust mite sublingual immunotherapy: a double-blind, placebo-controlled study in elderly patients with allergic rhinitis. Clin Exp Allergy. 2013 Feb;43(2):242-8. doi: 10.1111/cea.12039. PMID 23331565